CLINICAL TRIAL: NCT01123642
Title: Functional Outcomes in OEF/OIF Veterans With PTSD and Alcohol Misuse
Brief Title: Project SERVE: Post Deployment Functioning
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Texas A&M University (Other); Boston University (Other)
Responsible Party: Sponsor
Other Study IDs: D7202-R; 1I01RX000304-01A1 (NIH)
Record Dates: First submitted 2010-05-05; First posted 2010-05-14 (Estimated); Results first posted 2015-08-14 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Post-traumatic Stress Disorder; Depressive Disorder; Alcoholism
Keywords: post-traumatic stress disorder; depressive disorder; alcoholism; Longitudinal studies; readjustment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depressive Disorder; Alcoholism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Operation Enduring Freedom and Operation Iraqi Freedom Veterans

SUMMARY:
Functional recovery is of the utmost importance to evaluate in our returning Operation Enduring and Iraqi Freedom Veterans so that we can better understand their needs and experiences during the readjustment process from warzone to civilian life. Although most soldiers are resilient, concerning rates of PTSD (12-20%) and depression (14-15%) have been found, and as many as 24-35% report drinking more alcohol than they intended (Hoge et al., 2004). The current study proposes to follow returning Veterans for a one-year period to evaluate factors that influence the readjustment process and functional impairment. This information should guide the development of early intervention and treatment programs to help recovery.

DETAILED DESCRIPTION:
The proposed longitudinal study aims to better understand the functioning of returning Operation Enduring Freedom (OEF) and Operation Iraqi Freedom (OIF) OEF/OIF Veterans over time and to identify potentially malleable resilience factors associated with higher levels of functioning. A total of 300 returning OEF/OIF Veterans will be followed for a one-year period. Veterans will complete a baseline assessment, followed by three follow-up assessments (two self-report assessments mailed at 4- and 8-months post-baseline and a one-year in-person follow-up assessment that repeats many of the baseline clinician-administered assessments). Multiple functional outcomes will be evaluated, including occupational, family, social, and physical functioning. The specific aims include: 1) identifying whether a "dose-response" relationship exists between level of exposure to stressors (pre-deployment, deployment-related, and post-deployment) and functioning over time; 2) examining whether potentially malleable resilience factors predict higher levels of functioning in returning Veterans over time; 3) examining whether psychopathology predicts lower levels of functioning in returning Veterans over time; 4) testing the theoretical model that psychopathology partially mediates the effects of stress, social support, coping, and neurocognition on functioning over time; 5) examining whether changes in the use of healthy coping strategies, social support, post-deployment stress, and psychopathology predict changes in functioning over time; and 6) exploring whether stress, social support, coping, neurocognition, and psychopathology have differential effects on specific aspects of functioning (e.g., occupational, family, social, and physical functioning) over time. The long-term aim of this research is to develop evidence-based early intervention and treatment programs designed to assist returning OEF/OIF Veterans with achieving optimal functioning when reintegrating into civilian life. In keeping with the VHA's goal of operationalizing principles of recovery and rehabilitation in treatment planning, this research should provide a platform of empirical data to assist with the further development of meaningful early intervention and treatment programs to assist OEF/OIF Veterans with the post-war readjustment process over time.

ELIGIBILITY:
Inclusion Criteria:

To be eligible, participants must be:

* enrolled returning OEF/OIF Veteran within CTVHCS;
* English-speaking Veterans;
* able to comprehend and sign the informed consent form;
* able to complete the structured interviews and self-report assessments;
* willing to be contacted for follow-up assessments;
* deemed stable on psychotropic medications and in psychotherapy.

Exclusion Criteria:

Veterans will be excluded if they:

* plan to relocate out of the Central Texas area within four months of protocol initiation;
* meet criteria for a diagnoses of schizophrenia, other psychotic disorders, or bipolar disorder;
* report current hallucinations or delusions that are clearly not trauma-related; or
* report current suicidal or homicidal risk warranting crisis intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Operation Enduring Freedom and Operation Iraqi Freedom Veterans
Sampling Method: Non-Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2010-10; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra B Morissette, PhD, Principal Investigator — Central Texas Veterans Health Care System Waco VA Medical Center, Waco, TX
Locations (1):
- Central Texas Veterans Health Care System Waco VA Medical Center, Waco, TX, Waco, Texas, United States

REFERENCES:
- [Background] Dolan S, Martindale S, Robinson J, Kimbrel NA, Meyer EC, Kruse MI, Morissette SB, Young KA, Gulliver SB. Neuropsychological sequelae of PTSD and TBI following war deployment among OEF/OIF veterans. Neuropsychol Rev. 2012 Mar;22(1):21-34. doi: 10.1007/s11065-012-9190-5. Epub 2012 Feb 18. PMID 22350690
- [Background] Konecky B, Meyer EC, Marx BP, Kimbrel NA, Morissette SB. Using the WHODAS 2.0 to assess functional disability associated with DSM-5 mental disorders. Am J Psychiatry. 2014 Aug;171(8):818-20. doi: 10.1176/appi.ajp.2014.14050587. No abstract available. PMID 25082488
- [Result] Greenawalt DS, Tsan JY, Kimbrel NA, Meyer EC, Kruse MI, Tharp DF, Gulliver SB, Morissette SB. Mental Health Treatment Involvement and Religious Coping among African American, Hispanic, and White Veterans of the Wars of Iraq and Afghanistan. Depress Res Treat. 2011;2011:192186. doi: 10.1155/2011/192186. Epub 2011 Jul 18. PMID 21785719
- [Result] Morissette SB, Woodward M, Kimbrel NA, Meyer EC, Kruse MI, Dolan S, Gulliver SB. Deployment-related TBI, persistent postconcussive symptoms, PTSD, and depression in OEF/OIF veterans. Rehabil Psychol. 2011 Nov;56(4):340-50. doi: 10.1037/a0025462. PMID 22121940
- [Result] Debeer BB, Kimbrel NA, Meyer EC, Gulliver SB, Morissette SB. Combined PTSD and depressive symptoms interact with post-deployment social support to predict suicidal ideation in Operation Enduring Freedom and Operation Iraqi Freedom veterans. Psychiatry Res. 2014 May 30;216(3):357-62. doi: 10.1016/j.psychres.2014.02.010. Epub 2014 Feb 17. PMID 24612971
- [Result] Stock EM, Kimbrel NA, Meyer EC, Copeland LA, Monte R, Zeber JE, Gulliver SB, Morissette SB. A Bayesian model averaging approach to examining changes in quality of life among returning Iraq and Afghanistan veterans. Int J Methods Psychiatr Res. 2014 Sep;23(3):345-58. doi: 10.1002/mpr.1442. Epub 2014 Jun 18. PMID 24942672
- [Result] Grosso JA, Kimbrel NA, Dolan S, Meyer EC, Kruse MI, Gulliver SB, Morissette SB. A test of whether coping styles moderate the effect of PTSD symptoms on alcohol outcomes. J Trauma Stress. 2014 Aug;27(4):478-82. doi: 10.1002/jts.21943. PMID 25158641
- [Result] Kimbrel NA, Evans LD, Patel AB, Wilson LC, Meyer EC, Gulliver SB, Morissette SB. The critical warzone experiences (CWE) scale: initial psychometric properties and association with PTSD, anxiety, and depression. Psychiatry Res. 2014 Dec 30;220(3):1118-24. doi: 10.1016/j.psychres.2014.08.053. Epub 2014 Sep 6. PMID 25238984
- [Result] Kimbrel NA, Morissette SB, Meyer EC, Chrestman R, Jamroz R, Silvia PJ, Beckham JC, Young KA. Effect of the 5-HTTLPR polymorphism on posttraumatic stress disorder, depression, anxiety, and quality of life among Iraq and Afghanistan veterans. Anxiety Stress Coping. 2015;28(4):456-66. doi: 10.1080/10615806.2014.973862. Epub 2014 Nov 14. PMID 25314020
- [Result] Wilson LC, Kimbrel NA, Meyer EC, Young KA, Morissette SB. Do child abuse and maternal care interact to predict military sexual trauma? J Clin Psychol. 2015 Apr;71(4):378-86. doi: 10.1002/jclp.22143. Epub 2014 Dec 22. PMID 25534500
- [Result] Kimbrel NA, DeBeer BB, Meyer EC, Silvia PJ, Beckham JC, Young KA, Morissette SB. An examination of the broader effects of warzone experiences on returning Iraq/Afghanistan veterans' psychiatric health. Psychiatry Res. 2015 Mar 30;226(1):78-83. doi: 10.1016/j.psychres.2014.12.007. Epub 2014 Dec 13. PMID 25541538
- [Result] Hiraoka R, Meyer EC, Kimbrel NA, DeBeer BB, Gulliver SB, Morissette SB. Self-Compassion as a prospective predictor of PTSD symptom severity among trauma-exposed U.S. Iraq and Afghanistan war veterans. J Trauma Stress. 2015 Apr;28(2):127-33. doi: 10.1002/jts.21995. Epub 2015 Mar 21. PMID 25808565
- [Derived] Myers MN, Kurz AS, Paul J, Wild MG, O'Brien SF. Gender differences in reported potentially morally injurious events among post-9/11 U.S. combat veterans, using two measures. Psychol Trauma. 2025 Nov;17(8):1751-1761. doi: 10.1037/tra0001782. Epub 2024 Nov 7. PMID 39509229

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 345 participants were consented into the study, after which final eligibility was determined during the baseline assessment (see inclusion/exclusion criteria). Of the 345 enrolled, 309 met inclusion criteria and were deemed eligible for follow-up in the longitudinal study.
Groups:
- OEF/OIF/OND Veterans: Operations Enduring Freedom, Iraqi Freedom and New Dawn Veterans
Period: Overall Study
Arm/Group | OEF/OIF/OND Veterans
Started | 345
Completed | 277
Not Completed | 68
Not completed — Lost to Follow-up | 23
Not completed — Withdrawal by Subject | 9
Not completed — ineligible at baseline assessment | 36

BASELINE CHARACTERISTICS:
Population: A total of 345 participants were enrolled (signed informed consent), of which 309 met final eligibility criteria. Results are analyzed using the 309 eligible enrolled participants.
Arm/Group | OEF/OIF/OND Veterans
Number analyzed (Participants) | 309
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.81 (9.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 209

OUTCOME MEASURES:

1. Primary Outcome: World Health Organization Disability Assessment Schedule II (WHODAS II)
Description: Participants complete the WHODAS II at baseline, 4 months, 8 months, and 12 months. The WHODAS II measures general disability related to multiple domains (i.e., understanding and communicating, getting around, self care, getting along with people, life activities, work/school, participation in society). Total scores range from 1 (no disability) to 5 (extreme/cannot do), with higher scores indicating more impairment.
Time Frame: one year
Population: A total of 345 participants were enrolled, of which 309 were deemed eligible. Analyses are conducted with the total sample N = 309, followed over time. Sample sizes vary over time due to attrition and missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OEF/OIF/OND Veterans
Number analyzed (Participants) | 309
units on a scale
  Baseline: number analyzed (Participants) | 307
  Baseline | 1.87 (.69)
  4 months: number analyzed (Participants) | 266
  4 months | 2.03 (.77)
  8 months: number analyzed (Participants) | 256
  8 months | 2.07 (.78)
  12 months: number analyzed (Participants) | 254
  12 months | 1.88 (.73)

2. Secondary Outcome: Inventory of Psychosocial Functioning (IPF)
Description: 80-item self-report measure of psychosocial functioning across multiple domains (e.g., family, social, day-to-day activities). Items are rated on a 7-point scale ranging from 0 ("never") to 6 ("always"). Lower scores indicate more positive outcomes.
Time Frame: one year
Population: Sample sizes differ due to attrition and missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- OEF/OIF/OND Veterans: Operation Enduring Freedom/Operation Iraqi Freedom/Operation New Dawn Veterans
Arm/Group | OEF/OIF/OND Veterans
Number analyzed (Participants) | 305
score on a scale
  Baseline | 2.51 (1.25)
  12 months: number analyzed (Participants) | 268
  12 months | 2.33 (1.19)

3. Secondary Outcome: Quality of Life Scale (QLS)
Description: Quality of life measure of functioning scored on a 1 (delighted) to 7 (terrible) scale. Scores are summed with higher scores indicating lower quality of life. Total scores range from 16 - 112.
Time Frame: one year
Population: Sample sizes differ due to attrition and missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OEF/OIF/OND Veterans
Number analyzed (Participants) | 303
score on a scale
  Baseline | 76.33 (17.46)
  4 months: number analyzed (Participants) | 291
  4 months | 73.04 (20.20)
  8 months: number analyzed (Participants) | 272
  8 months | 72.38 (20.60)
  12 months: number analyzed (Participants) | 265
  12 months | 77.59 (18.31)

4. Secondary Outcome: Clinician Administered PTSD Scale (CAPS-5)
Description: Total scores reflecting PTSD symptom severity. Scores ranging from 0-136 (higher score = more severe).
Time Frame: one year
Population: Sample sizes differ across time points due to attrition and missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OEF/OIF/OND Veterans
Number analyzed (Participants) | 309
score on a scale
  Baseline | 29.71 (27.49)
  12 months: number analyzed (Participants) | 262
  12 months | 34.29 (30.94)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for a one year period (baseline to final assessment at 12 months).
Description: A total of 345 were enrolled, of which 309 were determined to be eligible. No adverse events occurred at the baseline assessment. Adverse events were reported with respect to the 309 eligible participants followed over time.
Arm/Group | OEF/OIF/OND Veterans
Serious Adverse Events (participants affected / at risk) | 28/309
Other Adverse Events (participants affected / at risk) | 2/309
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OEF/OIF/OND Veterans (N=309)
hospitalized for suicidal ideation/attempt (Psychiatric disorders) | 6
hospitalized for homicidal ideation (Psychiatric disorders) | 1
Hospitalized for mental health (Psychiatric disorders) | 3
Hospitalized for physical condition (General disorders) | 11
ER for physical condition (General disorders) | 7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OEF/OIF/OND Veterans (N=309)
Visit to ER for chest pain (Gastrointestinal disorders) | 1
Detained in jail (Social circumstances) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No